CLINICAL TRIAL: NCT01606527
Title: Prospective, Double-blind, Randomized, Placebo-controlled Trial of Ibuprofen Versus Placebo for Prevention of Neurologic Forms of Altitude Sickness
Brief Title: NSAID RCT for Prevention of Altitude Sickness
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Naval Health Research Center (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Gertsch MD, Senior Scientist, Warfighter Performance Laboratory, Naval Health Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NHRC.2012.0013
Record Dates: First submitted 2012-04-13; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Spectrum of Altitude-associated Neurologic Forms of Altitude
Keywords: Spectrum of Altitude-associated acute mountain sickness; hypoxia; high altitude headache; high altitude cerebral edemat is.....
MeSH Terms: conditions — Hypoxia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen 600mg taken three times daily for four days.
  Interventions: Drug: Ibuprofen 600mg orally three times daily
- placebo (Placebo Comparator): Avicel placebo capsules three times daily for four days
  Interventions: Drug: Ibuprofen 600mg orally three times daily

INTERVENTIONS:
Drug: Ibuprofen 600mg orally three times daily — Ibuprofen is taken 600mg orally three times daily
  Other Names: Motrin

SUMMARY:
The proposed study is a prospective, randomized, double-blind, placebo-controlled clinical trial evaluating ibuprofen and placebo for the prevention of neurological forms of altitude illness [including high altitude headache (HAH), acute mountain sickness (AMS), high altitude cerebral edema (HACE), and an emerging concept of High Altitude Anxiety]. The study will take place in the spring and summer of 2012 at the Marine Corps Mountain Warfare Training Center in the Eastern Sierras near Bridgeport, California. US Marines from near sea level will participate in battalion-level training exercises at between 8,500-11,500 Feet, where some altitude illness is expected. Concurrent measures used to determine objective markers of altitude illness, such that validated clinical scales, rapid cognitive screening tests, will inform us of symptoms of altitude illness.

ELIGIBILITY:
INCLUSION CRITERIA:

Active duty military

Current in their medical screening

EXCLUSION CRITERIA:

Upper respiratory tract infection or influenza

Have had a reaction to Ibuprofen, aspirin or other Non-Steroidal Anti-inflammatory Drugs (NSAIDs).

Stayed the night at an altitude of greater than 6,700 feet within the last 7 days

Headache at baseline

Have altitude sickness or more than one mild symptom of any severity on the Lake Louise Questionnaire including headache, poor appetite, nausea, vomiting, fatigue, weakness, dizziness, and/or poor sleep (insomnia)

Low blood oxygen or low oxygen saturation (<90%)

Pregnant or cannot exclude the possibility of being pregnant, or have missed menses by over 7 days.

Have taken any of the following in 48 hours preceding enrollment: acetazolamide/Diamox, steroids (dexamethasone/Decadron, prednisone), theophylline, or diuretics such as Lasix

Have taken any of the following within 12 hours preceding enrollment: Ibuprofen/Motrin, Naprosyn/Naproxen/Aleve, aspirin, or Acetaminophen/Tylenol.

Have taken any other medication that may be known to have potential for drug-drug interactions with ibuprofen, including (but not limited to): ACE-inhibitor antihypertiensives, thiazide diuretics, furosemide, lithium, methotrexate, and H-2 Agonists.

Have any medical conditions which may make participation hazardous (*by self-report which can be clarified before enrollment with the study physicians as necessary), including:

* Heart disease - Congestive heart failure, heart attack in the last month or severe coronary artery disease, or significant heart valve problems or other congenital problems.
* Lung disease - Restrictive lung disease, chronic obstructive pulmonary disease (COPD), severe obstructive sleep apnea, or pulmonary hypertension of any cause.
* Neurological disorders - Hydrocephalus, history of brain tumor, history of severe brain trauma or coma, pseudotumor cerebri, or severe uncontrolled headaches/migraine disorder (as diagnosed by a doctor).
* Gastrointestinal - Known stomach ulcer or history of gastrointestinal bleeding.
* Blood disorders - Anemia, leukemia, or other coagulopathies of any kind.
* Kidney disease - Kidney failure or other known kidney disease.

General - The Principal Investigator and co-investigator reserve the right to exclude a potential participant with conditions that in their judgment are not listed above, but which would reasonably represent concern for the participant's health and welfare, including (but not limited to) conditions that may directly antagonize mechanisms of acclimatization to altitude, organ failure, metastatic/malignant neoplasm, space-occupying brain lesions or diagnoses typically known to raise intracranial pressure, and disorders that are likely to antagonize adequate respiration, blood oxygenation, and/or circulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of AMS as measured on the Lake Louise AMS Questionnaire across the study. | Twice daily
  The measure is assessed twice daily for four days

SECONDARY OUTCOMES:
1. Change in High Altitude Headache measured by the Visual Analog Scale (VAS) across the study. | Twice daily
  The measure is assessed twice daily for four days
2. Change in cognitive performance as measured by King-Devick across the study. | Twice daily
  The measure is assessed twice daily for four days
3. Change in the presence of anxiety and somatic symptoms using the BSI-12 screening tool across the study | Twice daily
  The measure is assessed twice daily for four days
4. Change in the oxygen concentration using Pulse Oximetry across the study. | Twice daily
  The measure is assessed twice daily for four days
5. Change in hydration status as measured by urine specific gravity across the study. | Twice daily
  The measure is assessed twice daily for four days
6. Change in HAH incidence and severity as measured on the Lake Louise AMS Questionnaire across the study. | Twice daily
  The measure is assessed daily for four days
7. Change in cognitive performance as measured by the Quickstick across the study | Twice daily
  The measure is assessed twice daily for four days
8. Change in the presence of anxiety and somatic symptoms using the GAD-2 screening tool across the study | Twice daily
  The measure is assesed twice daily for four days
9. Incidence of severe AMS as measured by a score of 6 or greater on the Lake Louise AMS Questionnaire. | Twice Daily
  The measure is assessed twice daily for four days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Gertsch, MD, Principal Investigator — Naval Health Research Center - San Diego
Locations (1):
- Marine Mountain Warfare Training Center, Bridgeport, California, United States